CLINICAL TRIAL: NCT01763554
Title: Review of Medical Records of Patients Who Have Been Treated With Lutetium at the Cross Cancer Institute Between January 2010 and April 30, 2014
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: REV-LUT-001
Record Dates: First submitted 2012-12-19; First posted 2013-01-09 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Neuroendocrine Tumors, NET
Keywords: Lu-177; Lutetium-177; DOTA-TATE; Neuroendocrine tumors; radiopharmaceutical
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lu-177 DOTA-TATE — The regimen used for therapy for patients treated under SAP was a standard dose of 5.55 GBq Lu-177 DOTA-TATE every 10-12 weeks for 4 treatments, then every 6 months as maintenance treatment.

SUMMARY:
Retrospective review of the medical files of 115 patients with neuroendocrine tumours who were treated with Lutetium-177 DOTA-TATE under Health Canada's Special Access Programme (SAP) at the Cross Cancer Institute between January 2010 and April 30, 2014. Efficacy, safety, and other relevant data will be collected to support a separate clinical trial application.

ELIGIBILITY:
Subjects with neuroendocrine tumours who received Lu-177 DOTA-TATE treatment under SAP at the Cross Cancer Institute between January 2010 and April 30, 2014.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Limited to those subjects with neuroendocrine tumors who received Lu-177 DOTA-TATE treatment under SAP at the Cross Cancer Institute between January 2010 and April 30, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2012-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy data on subjects with neuroendocrine tumours (NET) treated with Lu-177 DOTA-TATE | Retrospective data January 2010 - April 30, 2014
  Data (Radioisotope and CT/MRI images, blood assays and Quality of Life Questionnaires, pre and post treatment) will be collected to determine tumor response of subjects with NET after treatment with Lu-177 DOTA-TATE.

SECONDARY OUTCOMES:
Safety and other relevant information on subjects treated with Lu-177 DOTA-TATE | Retrospective data January 2010 - April 30, 2014
  Safety data will include blood counts and chemistry, GFR and adverse events, pre and post treatment. Other data includes patient demographics.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Morrish, MD, PhD, Principal Investigator — Endocrinology & Oncology, University of Alberta, Cross Cancer Institute
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada